CLINICAL TRIAL: NCT02109068
Title: Lifestyle, Exercise and Nutrition (LEAN) Study 1
Brief Title: Lifestyle, Exercise and Nutrition Study 1
Acronym: LEAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1012007780
Record Dates: First submitted 2014-04-04; First posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer; Weight Loss
Keywords: Breast Cancer; Survivorship; Weight Loss
MeSH Terms: conditions — Breast Neoplasms; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- In-Person Counseling (Active Comparator): Participants randomized to in-person counseling will meet via in-person or via telephone (but at least 3 of the 11 sessions must be in person) weekly for month 1, then every other week for months 2, and 3, and then monthly for months 4-6 at Yale University. The meetings will last 30 minutes. Participants will turn in their diet and exercise logs and also be weighed. A lesson will then be discussed (see above for content).
  Interventions: Behavioral: Weight Loss Counseling- In-Person
- Telephone-based Counseling (Active Comparator): The exact same information, content, schedule, and 30 minute sessions will be provided to telephone-based participants as offered to participants who receive in-person counseling. Participants will be taught diet, exercise and behavior change strategies via the telephone (weekly calls for month 1, every other week for months 2-3, and monthly for months 4-6). All lessons and diet and physical activity logs will be mailed to them at the beginning of the program. Participants will record their daily diet and exercise in the logs. Every four weeks, participants will return, via stamped, addressed envelopes, the logs to the study office.
  Interventions: Behavioral: Weight Loss Counseling- Phone
- Usual Care (No Intervention): Immediately after randomization, participants in the Usual Care Group will be provided written information that emphasizes the importance of a healthy lifestyle. Usual care participants will be encouraged to follow the American Cancer Society (ACS) nutrition and physical activity guidelines. Upon completion of the study (at 6 months), usual care participants will be offered all the educational material, as well as an in-person or telephone counseling session.

INTERVENTIONS:
Behavioral: Weight Loss Counseling- Phone — The intervention will be based on the Diabetes Prevention Program weight loss program, which uses a combination of reduced caloric intake, increased physical activity, and behavior therapy. The content of the weight loss program will be similar for the in-person and telephone interventions, but the approach will vary (i.e., in-person vs. telephone counseling). The weight loss intervention will be conducted by a Registered Dietitian, who has training in exercise physiology and behavior modification.
  During the 6-month intervention, participants will receive weekly (month 1), then bi-weekly (months 2 and 3), then monthly (months 4, 5, and 6) individualized counseling sessions. An advantage of tapering the frequency of visits from weekly to every other week and then monthly works as a process tool to help transfer the work or responsibility onto the participant for life long change and maintenance of behavior change.
  Arms: Telephone-based Counseling
Behavioral: Weight Loss Counseling- In-Person — The intervention will be based on the Diabetes Prevention Program weight loss program, which uses a combination of reduced caloric intake, increased physical activity, and behavior therapy. The content of the weight loss program will be similar for the in-person and telephone interventions, but the approach will vary (i.e., in-person vs. telephone counseling). The weight loss intervention will be conducted by a Registered Dietitian, who has training in exercise physiology and behavior modification.
  During the 6-month intervention, participants will receive weekly (month 1), then bi-weekly (months 2 and 3), then monthly (months 4, 5, and 6) individualized counseling sessions. An advantage of tapering the frequency of visits from weekly to every other week and then monthly works as a process tool to help transfer the work or responsibility onto the participant for life long change and maintenance of behavior change.
  Arms: In-Person Counseling

SUMMARY:
The specific aims of this study are to determine the efficacy and cost-effectiveness of a weight loss program compared with usual care (control) treatment on 6-month changes in body weight, body fat, and serum hormones in breast cancer survivors.

DETAILED DESCRIPTION:
Proposed is a three-arm randomized controlled trial of 6-months of weight loss counseling (i.e., dietary-induced caloric restriction and physical activity) on clinically meaningful endpoints in 100 breast cancer survivors . The three arms will be: 1. In-person counseling, 2. Telephone-based counseling, 3. Usual care. Women will be randomized into one of 3 study arms using a random permuted block design. Research staff collecting body composition data, as well as reviewing forms and entering data, will be blinded to the participant's study group.

ELIGIBILITY:
Inclusion Criteria:

* American Joint Committee on Cancer (AJCC) Stages 0-IIIC Breast Cancer
* BMI >25 kg/m2
* Completed surgery, chemotherapy and radiation at least 2 months ago
* Physically able to exercise
* Agrees to be randomly assigned to either weight loss or control
* Gives informed consent to participate in all study activities
* Able to come for baseline and 6-month clinic visits
* Mentally competent

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | 6 months
  BMI will be calculated using weight and height measurements (weight (kg)/height (m)^2 ). Weight and height will be measured by research staff blinded to the participant's randomization group at baseline and 6-months. Participants will be weighed in light indoor clothing, without shoes, rounding up to the nearest 0.1 kg; height will be measured in a standard manner, without shoes, using a stadiometer, rounding up to the nearest 0.1 cm. All measures will be performed and recorded twice in succession.
Change in body weight in kilograms (kg) | 6 months
  Participants will be weighed in light indoor clothing, without shoes, rounding up to the nearest 0.1 kg. All measures will be performed and recorded twice in succession.
Change in percent body fat | 6 months
  Dual Energy X-Ray Absorptiometry (DEXA) scans will be performed at baseline and 6-months. The DEXA measurements will be made with a Hologic scanner (Hologic 4500 with a "Discovery" upgrade, Hologic Inc, Waltham, Mass). A whole-body scan takes approximately 10 minutes to complete. Percent body fat will be measured utilizing DEXA.

SECONDARY OUTCOMES:
Change in fasting insulin | 6 months
  All the hormones to be measured (insulin, IGF-1, leptin, adiponectin and C-reactive protein) have been previously measured in our lab and published. Immunoassay techniques and kits from Diagnostic Products Corporation (DPC, Los Angeles, CA) to will be used to measure each hormone value. Each woman's baseline and follow-up samples will be used in the same batch, and an equal number of intervention and control samples will also be included in the same batch. Blind duplicates are also included in and between batches to estimate coefficient of variations.
Change in Insulin-like growth factor 1 (IGF-1) | 6 months
  All the hormones to be measured (insulin, IGF-1, leptin, adiponectin and C-reactive protein) have been previously measured in our lab and published. Immunoassay techniques and kits from Diagnostic Products Corporation (DPC, Los Angeles, CA) to will be used to measure each hormone value. Each woman's baseline and follow-up samples will be used in the same batch, and an equal number of intervention and control samples will also be included in the same batch. Blind duplicates are also included in and between batches to estimate coefficient of variations.
Change in Leptin | 6 months
  All the hormones to be measured (insulin, IGF-1, leptin, adiponectin and C-reactive protein) have been previously measured in our lab and published. Immunoassay techniques and kits from Diagnostic Products Corporation (DPC, Los Angeles, CA) to will be used to measure each hormone value. Each woman's baseline and follow-up samples will be used in the same batch, and an equal number of intervention and control samples will also be included in the same batch. Blind duplicates are also included in and between batches to estimate coefficient of variations.
Change in C-reactive protein | 6 months
  All the hormones to be measured (insulin, IGF-1, leptin, adiponectin and C-reactive protein) have been previously measured in our lab and published. Immunoassay techniques and kits from Diagnostic Products Corporation (DPC, Los Angeles, CA) to will be used to measure each hormone value. Each woman's baseline and follow-up samples will be used in the same batch, and an equal number of intervention and control samples will also be included in the same batch. Blind duplicates are also included in and between batches to estimate coefficient of variations.
Skin Carotenoids Assessment | 6 months
  Assessment of skin carotenoids will be done using Resonance RAMAN Spectroscopy (RRS). Briefly, a small scanner which shines blue light is placed on the palm of the hand for 30 seconds. The palm is cleaned with an alcohol wipe prior to the scan, A RRS reading is available after a further 30 seconds. The procedure is repeated at the same body location. Skin color is self assessed by the participants at the baseline visit using samples that are used in plastic surgery to assess skin color. Melanin content (skin color) may have a small effect on RRS, but this effect is minimized by assessing skin carotenoids in the palm, which has a lower melanin content than other body sites.
Maintenance of Weight Loss | 12 months
  A mailed follow up will be conducted at 12-months post randomization. Questionnaires will be mailed to the participant with a pre-paid envelope for their return. Information about current weight will be conducted using this method.

OTHER OUTCOMES:
Change in Physical Activity | 6 months
  The 7-Day Daily Activity Log (7-Day DAL) will be the primary measure used to compare physical activity levels at baseline and 6-months among the three groups. All participants will complete the log for seven consecutive days, recording the amount of time spent in moderate- to vigorous-intensity recreational exercise. Total minutes per week of exercise will be calculated. Participants randomized to in-person and telephone counseling will also complete the 7-day DAL weekly.
Change in Dietary Intake | 6 months
  The endpoint measures of diet change will be mean, group level changes in daily caloric intake, based on a 120-item food frequency questionnaire (FFQ) which was developed for the Women's Health Initiative Study and has been validated against 4-Day Food Records and 24-hour Dietary Recalls. FFQs will be administered at baseline and 6-months.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda L Irwin, PhD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States